CLINICAL TRIAL: NCT01752361
Title: Gastrointestinal Transit Times and Motility in Patients Suffering From Severe Ulcerative Colitis Obtained by Motilis-3D-transit
Brief Title: Gastrointestinal Transit Times and Motility in Severe Ulcerative Colitis Obtained by Motilis-3D-transit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Motilis Medica A/S ,Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: M-20110276
Record Dates: First submitted 2012-11-27; First posted 2012-12-19 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Ulcerative Colitis
Keywords: Gastrointestinal Motility; Inflammatory Bowel Disease; Transit time
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ulcerative Colitis
  Interventions: Device: Motilis-3D transit

INTERVENTIONS:
Device: Motilis-3D transit

SUMMARY:
The purpose of this study is to describe gastrointestinal (GI) motility in patients suffering from severe Ulcerative Colitis (UC) and to compare these results with similar results from a study on healthy subjects.

Both studies are done with the use of Motilis 3D-Transit system which consists of a small electronic capsule ingested and detected by a receiver carried by the patient. Position and orientation of the capsule are interpreted by dedicated computer software and transit times, progression velocity and contraction frequencies can be revealed.

The study is mainly descriptive and is designed to test and evaluate the usefulness of the Motilis 3D Transit system in UC patients and to tell us more about GI motility during severe inflammation.

Motilis 3D-Transit system gives us a unique chance to study the gastrointestinal canal as a whole during severe illness.

We expect to include 20 patients suffering from severe UC admitted to Hospital with the purpose of getting medical treatment. We do not expect any drop out, but in case of drop out a new patient will be included.

ELIGIBILITY:
Inclusion Criteria:

* Severe Ulcerative colitis (modified Truelove and Witt score)
* Signed informed consent obtained
* Fasted since midnight

Exclusion Criteria:

* Known GI related symptoms complaints or GI diseases
* Swallowing disorders
* Cancer or other life threatening diseases or conditions
* Pregnancy or breast-feeding
* Previous abdominal surgery
* Abdominal diameter >140cm?
* Drug abuse or alcoholism
* Irregular bowel movements
* Known cardiovascular or pulmonary diseases
* Participation in any clinical study within the last 30 days
* Cardiac pacemaker or infusion pump or any other implanted or portable electro-mechanical medical device.
* Medication affecting GI motility
* MRI within the next four weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe Ulcerative Colitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Velocity of progression through the inflamed part of the colon in severe UC compared to the velocity of progression in the corresponding colonic segment in healthy volunteers. | Three days from baseline visit

SECONDARY OUTCOMES:
Velocity of progression through the non-inflamed colonic segments in severe UC compared to the velocity of progression in the corresponding colonic segments in healthy volunteers. | Three days from baseline

OTHER OUTCOMES:
Velocity of progression through the small intestine in severe UC compared to velocity of progression through the small intestine in healthy volunteers. | three days from baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: AnneMette Haase, Ph.d Student, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Hepato and Gastroenterolegy, Aarhus C, Denmark